CLINICAL TRIAL: NCT01242852
Title: SIGnificance of Routine Hysteroscopy Prior to a First 'in Vitro Fertilization'(IVF) Treatment Cycle
Acronym: inSIGHT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Erasmus Medical Center (Other); Maastricht University Medical Center (Other); Maxima Medical Center (Other)
Responsible Party: Principal Investigator, Bart CJM Fauser, MD, PhD, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: inSIGHT
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Intrauterine Abnormalities in Infertility
Keywords: Hysteroscopy; infertility; subfertility; intrauterine abnormalities; intracavitary pathology; IVF; ICSI; in vitro fertilization; intracytoplasmic sperm injection
MeSH Terms: conditions — Infertility | interventions — Hysteroscopy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Additional diagnostic tests (Experimental): Participants in the experimental arm will undergo standard hysteroscopy with treatment-on-the spot of predefined intrauterine abnormalities. In two of the participating clinics, also a 'Saline Infusion Sonography' (SIS) will be performed, 1 week before the hysteroscopy. After the additional diagnostic test(s), standard IVF/ICSI treatment will be initiated.
  Interventions: Procedure: Office hysteroscopy (in combination with a 'Saline Infusion Sonography'(SIS))
- Routine fertility workup (No Intervention): Patients allocated to the conventional strategy will be scheduled for IVF and undergo standard treatment, without SIS or hysteroscopy.

INTERVENTIONS:
Procedure: Office hysteroscopy (in combination with a 'Saline Infusion Sonography'(SIS)) — Routine fertility work-up, added up with diagnostic tests. In 5 research centers the extra tests consist of SIS & hysteroscopy (HY). In the other research hospitals it consists of only a HY. The HY examination will be scheduled on Day 3-12 of a cycle. It will be performed in an outpatient setting with a vaginoscopic approach. A 5-mm diameter continuous flow hysteroscope and a 30º direction of view will be used. The uterus will be inspected methodically a endometrial biopsy obtained and the findings recorded into a standardized form. Intrauterine pathology is defined as septum, endometrial polyp, submucous myoma, adhesions & endometritis. These will be treated, using scissors, Versapoint, grasping forceps, polyp snare or antibiotics. In 5 of the research hospitals, 1 week prior to the HY, also a SIS will be performed. Via a catheter saline solution will be infused into the uterine cavity as distention media. The findings at the following sonography will be standardized recorded.
  Other Names: Hysteroscopy
  Arms: Additional diagnostic tests

SUMMARY:
BACKGROUND: Despite the numerous advances in the field of in vitro fertilisation/intracytoplasmic sperm injection (IVF/ICSI), there still exists a maximum implantation rate per embryo transferred of about 30%. Next to the physiological and physic burden that comes with every IVF treatment cycle, implantation failure also adds up to the considerable costs associated with ART. Studies have shown, that minor intrauterine abnormalities can be found in 11-40% of the infertile women with a normal transvaginal sonography. Detection and treatment of these abnormalities by office hysteroscopy have led to a 9-13% increase in pregnancy rate. Therefore, it is increasingly advocated to screen all infertile women on intracavitary pathology prior to the start of IVF/ICSI.

OBJECTIVE: The aim of the proposed study is to assess whether diagnosing and treating unsuspected intrauterine abnormalities by saline infusion sonography and/or routine office hysteroscopy prior to a first IVF/ICSI treatment cycle improves the cost-effectiveness of the fertility treatment.

STUDY DESIGN: Multicenter randomized intervention study. POPULATION: Asymptomatic women, indicated for a first IVF/ICSI treatment cycle and a normal transvaginal ultrasonography.

INTERVENTION: Participants will be randomized for a (SIS and) hysteroscopy with treatment-on-the spot of predefined intrauterine abnormalities versus no diagnostic work-up. In both groups standard IVF/ICSI treatment will be initiated.

PRIMARY OUTCOME MEASURE:

Cumulative ongoing pregnancy rate resulting in live birth achieved within 18 months of IVF/ICSI treatment after randomization (obtained in both treatment cycles with fresh embryos, as well as in subsequent cryo/thaw cycles)

SECONDARY OUTCOME MEASURE:

* Cumulative implantation rate achieved within 18 months of IVF/ICSI treatment after randomization (obtained in both treatment cycles with fresh embryos, as well as in subsequent cryo/thaw cycles)
* Cumulative miscarry rate within 18 months of IVF/ICSI treatment after randomization (obtained in both treatment cycles with fresh embryos, as well as in subsequent cryo/thaw cycles)
* Cost calculations of, SIS, hysteroscopy procedures and the IVF treatment
* Patient preference and tolerance of a SIS and diagnostic/therapeutic hysteroscopy procedure
* Prevalence of unexpected intrauterine abnormalities
* Diagnostic accuracy of SIS in diagnosing intrauterine abnormalities

ELIGIBILITY:
Inclusion Criteria:

* Women indicated for a first IVF/ICSI treatment
* Primary or secondary infertility
* Normal Transvaginal Ultrasound, performed in the follicular phase of the menstrual cycle

Exclusion Criteria:

* Recurrent miscarriage
* Prior hysteroscopy treatments
* Meno-metrorrhagia (defined as any intermenstrual loss of blood)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2011-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy | 18 months
  Cumulative ongoing pregnancy rate resulting in live birth achieved within 18 months of IVF/ICSI treatment after randomisation (obtained in both treatment cycles with fresh embryos, as well as in subsequent cryo/thaw cycles)

SECONDARY OUTCOMES:
Implantation rate | 18 months
  Cumulative implantation rate achieved within 18 months of IVF/ICSI treatment after randomisation (obtained in both treatment cycles with fresh embryos, as well as in subsequent cryo/thaw cycles)
Miscarry rate | 18 months
  Cumulative miscarry rate within 18 months of IVF/ICSI treatment after randomisation (obtained in both treatment cycles with fresh embryos, as well as in subsequent cryo/thaw cycles)
Costs | 24 months
  Cost calculations of, SIS, hysteroscopy procedures and the IVF treatment
Patient tolerance | 24 months
  Patient tolerance of a SIS and diagnostic/therapeutic hysteroscopy procedure
Prevalence of unexpected intrauterine abnormalities | 3 months
Diagnostic accuracy of SIS | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Smit JG, Kasius JC, Eijkemans MJC, Koks CAM, van Golde R, Nap AW, Scheffer GJ, Manger PAP, Hoek A, Schoot BC, van Heusden AM, Kuchenbecker WKH, Perquin DAM, Fleischer K, Kaaijk EM, Sluijmer A, Friederich J, Dykgraaf RHM, van Hooff M, Louwe LA, Kwee J, de Koning CH, Janssen ICAH, Mol F, Mol BWJ, Broekmans FJM, Torrance HL. Hysteroscopy before in-vitro fertilisation (inSIGHT): a multicentre, randomised controlled trial. Lancet. 2016 Jun 25;387(10038):2622-2629. doi: 10.1016/S0140-6736(16)00231-2. Epub 2016 Apr 27. PMID 27132052
- [Derived] Smit JG, Kasius JC, Eijkemans MJ, Koks CA, Van Golde R, Oosterhuis JG, Nap AW, Scheffer GJ, Manger PA, Hoek A, Kaplan M, Schoot DB, van Heusden AM, Kuchenbecker WK, Perquin DA, Fleischer K, Kaaijk EM, Sluijmer A, Friederich J, Laven JS, van Hooff M, Louwe LA, Kwee J, Boomgaard JJ, de Koning CH, Janssen IC, Mol F, Mol BW, Torrance HL, Broekmans FJ. The inSIGHT study: costs and effects of routine hysteroscopy prior to a first IVF treatment cycle. A randomised controlled trial. BMC Womens Health. 2012 Aug 8;12:22. doi: 10.1186/1472-6874-12-22. PMID 22873367
- See also: All consortium studies performed multicentered in The Netherlands — http://www.studies-obsgyn.nl/